CLINICAL TRIAL: NCT05705271
Title: A Prospective, Interventional, Multicenter, Phase IV, Open-label, Single Arm Study to Assess the Safety and Effectiveness of Finerenone in Participants From India With Chronic Kidney Disease Associated With Type 2 Diabetes.
Brief Title: A Study to Learn How Safe the Study Drug Finerenone is and How Well it Works in Indian People With Long-term Decrease in the Kidneys' Ability to Work Properly (Chronic Kidney Disease) Together With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22224
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — finerenone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Finerenone (Experimental): Participants will receive study treatment for 18 months ± 7 days.
  Interventions: Drug: Finerenone (Kerendia, BAY94-8862)

INTERVENTIONS:
Drug: Finerenone (Kerendia, BAY94-8862) — Film-coated tablet, oral administration, once daily (OD), dosage based on the eGFR and serum potassium thresholds

SUMMARY:
Researchers are looking for a better way to treat people with chronic kidney disease (CKD), a progressive decrease in the kidneys' ability to work properly, and type 2 diabetes (T2D).

In people with T2D, the body does not make enough of a hormone called insulin or does not use the insulin well enough. Insulin's role is to regulate the amount of glucose (sugar) in the blood. Too much blood sugar can cause damage to the kidneys over time. Consequently, CKD can happen as one of the complications of T2D.

The study treatment finerenone works by blocking a group of proteins, called mineralocorticoid receptor. An increased stimulation of the mineralocorticoid receptor is known to trigger injury and inflammation in the kidney and is therefore thought to play a role in CKD.

Finerenone is already available in several countries for doctors to prescribe to people with CKD and T2D. In addition, it was recently approved in India with a request to specifically gather information on finerenone therapy in Indians.

The main purpose of this study is to learn how safe finerenone is in Indian people with CKD and T2D. For this, the researchers will count the number of participants who have:

* medical problems after taking finerenone
* abnormal high levels of potassium in the blood (called hyperkalemia).

Researcher will also count the number of participants in whom hyperkalemia:

* leads to stop of finerenone treatment
* requires treatment to filter wastes and water from the blood
* leads to a hospital stay.

Doctors keep track of all medical problems that happen in studies, even if they do not think the medical problems might be related to the study treatments.

In addition, the study team will collect more data about how well finerenone works in Indian people with CKD and T2D under real world setting. Working well means that the treatment can prevent the following from happening:

* reduced kidney function over a period of at least 4 weeks
* death from renal problems
* death due to conditions affecting the heart and blood circulation
* heart attack (blocked blood flow to the heart)
* hospital stay due to a condition which occurs when the heart does not pump blood as well as it should
* changes of the albumin and creatinine levels in urine.

The participants will be in the study for approximately 20 months. They will take the study treatment once daily as a tablet by mouth for 18 months. In the study, 9 visits to the study site are planned.

During the study, the study team will:

* take blood and urine samples
* do physical examinations
* check the participants' overall health
* do pregnancy tests
* examine heart health using electrocardiogram ECG
* check vital signs.

About 30 days after the participants take their last treatment, the study doctors and their team will check worsening of reported underlying diseases:

* damage to the blood vessels in the tissue of the retina at the back of the eye, as a result of diabetes mellitus
* a long-term condition where the heart does not pump blood as well as it should with symptoms such as shortness of breath, tiredness and ankle swelling
* heart attack (blocked blood flow to the heart)
* death due to conditions affecting the heart and blood circulation or
* hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Participants capable of giving signed informed consent signed before any study-specific procedure and willing to comply with the study-related procedures.
* Diagnosis of chronic kidney disease (CKD) associated with type 2 diabetes (T2D).
* Participants who are drug naïve for finerenone or patients who have been initiated on finerenone therapy within 4 weeks before signing the informed consent.
* Participants with serum potassium level ≤ 4.8 mmol/L at the time of Screening. If serum potassium level > 4.8 to 5.0 mmol/L, participants may be enrolled in the study, but additional potassium samples may be required; the potassium level needs to be confirmed during Screening. Participants with potassium level > 5.0 mmol/L are not allowed. The sample for potassium assessment for confirming eligibility shall be available before initiation of treatment with finerenone.
* Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Contraindications according to the local marketing authorization:

  1. Participants with eGFR < 25 mL/min/1.73 m^2 (calculated based on the CKD-EPI equation, using 2009 formula). eGFR can be reassessed once within 48 hours.
  2. Participants with severe hepatic impairment (Child-Pugh C).
  3. Participants with known hypersensitivity to the study treatment (active substance or excipients).
  4. Participants with Type 1 Diabetes.
  5. Participants taking concomitant medications that are strong CYP3A4 inhibitors.
  6. Participants with Addison's disease.
* Glycated hemoglobin > 12% (17.5 mmol/L) at the Screening visit.
* Participants treated with another mineralocorticoid receptor antagonist (MRA), a renin inhibitor, potassium supplements, a potassium sparing diuretic, a potassium binder agent, or angiotensin receptor neprilysin inhibitor (ARNI) within 8 weeks prior to the Screening visit and during finerenone treatment.
* Participation in another interventional clinical trial within 30 days prior to the Screening visit and during finerenone treatment.
* Female participants who are pregnant or breast-feeding or plan to become pregnant or to breastfeed during the course of the study.
* Participants known for lack of compliance with clinic visits or prescribed medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (TESAEs) | From the first finerenone treatment date up to 30 days after the last treatment date
Number of participants with hyperkalemia events | Up to 19 months
  including hyperkalemia (serum potassium > 5.5 mmol/L), severe hyperkalemia (serum potassium > 6.0 mmol/L), hyperkalemia leading to study drug discontinuation, hyperkalemia leading to dialysis and hyperkalemia leading to hospitalization

SECONDARY OUTCOMES:
Time to the first occurrence of the composite of kidney failure, a sustained decrease of at least 40% in the estimated glomerular filtration Rate (eGFR) from baseline over a period of at least 4 weeks, or death from renal cause | Up to 19 months
Time to the first occurrence of composite of cardiovascular (CV) death, nonfatal myocardial infarction, or hospitalization for heart failure (HF) | Up to 19 months
Change in urine albumin-to-creatinine ratio (UACR) from baseline to 4 months | From baseline to 4 months

CONTACTS AND LOCATIONS:
Locations (17):
- India (17):
  - Bhate Hospital, Karnataka, Belagavi
  - Muljibhai Patel Urological Hospital (MPUH) (Kidney Hospital), Nadiād, Gujarat
  - Accord Superspeciality Hospital, Faridabad, Haryana
  - Kempegowda Institute of Medical Sciences Hospital & R C, Bangalore, Karnataka
  - Christian Medical College, Vellore, Kerala
  - Global Hospital-Super Speciality And Transplant Centre, Mumbai, Maharashtra
  - Lancelot Medical Centre, Mumbai, Maharashtra
  - Dr Balabhai Nanavati Hospital, Mumbai, Maharashtra,, Maharashtra
  - PSRI Institute of Renal Sciences, New Delhi, National Capital Territory of Delhi
  - Vardhman Mahavir Medical College & Safdarjung Hospital (VMMC-SJH), New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, Bhubaneswar, Odisha
  - Jawaharlal Institute Of Postgraduate Medical Education and R, Gorimedu, Puducherry
  - Government Stanley Medical College and Hospital, Chennai, Tamil Nadu
  - M.V. Hospital & Research Centre 314/30, Chowk Lucknow, Uttar Pradesh
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS), Lucknow, Uttar Pradesh
  - Medica Superspecialty Hospital, Kolkata, West Bengal
  - Nizam's Institute of Medical Sciences (NIMS), Hyderabad

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.